CLINICAL TRIAL: NCT05128149
Title: Metabolic Control and Patient Well-being in Phenylketonuria: do Guidelines Make a Difference?
Acronym: PKU_Guide
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: UChildrenVienna (Unknown); University Children's Hospital Basel (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: PKU_Guide
Record Dates: First submitted 2021-09-22; First posted 2021-11-19 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Treatment of PKU implies for most patients that with strict adherence to dietary treatment they can achieve excellent neurocognitive outcome. Dietary treatment, though, is hard to comply to every day and with every single meal. Unsurprisingly, health-related quality of life (HrQol) is negatively affected if patients have to follow a dietary regime of this kind. Adherence to treatment in PKU is very variable. Factors of significant impact on adherence to treatment and well-being in chronic disease such as self-efficacy or parenting stress have not yet been widely investigated in PKU patients.

The ideal treatment prescription (and guideline) recommends as much as necessary and as little as possible, based on the best evidence available. Patients should neither be deprived of treatment options nor be exposed to overtreatment.

This study investigates adherence, metabolic control, HrQol in PKU patients treated by centres which follow different guidelines

ELIGIBILITY:
Inclusion Criteria:- Patients with PKU from age 10 years requiring dietary and / or pharmacological treatment according to locally applied guidelines

* Parents of patients with PKU aged 10 to 18 years requiring dietary and / or pharmacological treatment according to locally applied guidelines
* Ability and willingness to answer the questionnaires and follow the study procedures
* Informed consent as documented by signature

Exclusion criteria for patients and parents :

* Inability to follow the procedures of the study, e.g. due to language problems or severely reduced health status
* Pregnant patients or patients who have disclosed to their physician that they are planning a pregnancy in the near future
* Hyperphenylalaninaemia or mild forms of PKU or other inborn errors associated with elevated Phe but not requiring dietary and / or pharmacological treatment according to locally applied guidelines
* No inform

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PKU patients > 10 years and their parents
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Phe values | report on measurements from past 24 months
  biochemical marker for PKU

SECONDARY OUTCOMES:
Health-related quality of life | one hour
  PKU-QoL© Questionnaire
Self-efficacy | one hour
  10 items Self-efficacy scale (Schwarzer& Jerusalem)
Burden on family (patients from 10-18 years) | one hour
  Revised Impact on Family Scale

CONTACTS AND LOCATIONS:
Locations (1):
- University Childrens Hospital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No